



## **Evaluating the Efficacy of Obturator Cryoneurotomy for Hip Adductor Spasticity**

NCT Number: Date: September 10,2021





# ASSENT FORM Hip Adductor Cryoneurotomy

#### Invitation

I am being invited to be a part of a research study. This study is going to help find the best treatments for kids like me. Whether or not I choose to be a part of the study will not affect how my doctors treat me. I do not have to be a part of the study if I do not want to. Nobody will be mad at me if I do not want to be in the study. Even if I agree to be in the study now, I can change my mind later.

#### Why Are We Doing This Study?

This study will help us learn more about cryoneurotomy. During cryoneurotomy, the doctor freezes a nerve with a cold needle. Freezing the nerve lets the tight muscles relax and makes it easier for people to move. It is being tested for children like me who have tight muscles on the inside of their thighs. This is called spasticity. Children who have spasticity like mine often have a hard time walking, playing, washing, and standing. I am being invited to be a part of the study because my doctor has decided to use cryoneurotomy to help with my spasticity.

#### What Will Happen in This Study?

If I agree to be in this study, I will only have to go to my normal appointments. I will do all of my normal tests and measurements. I will also do a test where the doctors take a video and time me walking ten meters. Nobody will be able to recognize me in the video. I will answer some quick questions about my pain. Doctors will look at my measurements and test results to see how they are changing.

#### Who Is Doing This Study?

**Dr. Paul Winston** and his team from Victoria General Hospital will be doing this study. They will answer any questions I have about the study. I can also call them at **250-727-4221** if I am having any problems or if there is an emergency and I cannot talk to my parents.

#### Can Anything Bad Happen to Me?





There is nothing in this study that will make anything bad happen to me. Steps are being taken prevent me from catching COVID-19 during my visits. Everybody in the clinic will be wearing masks. Everybody who works in the clinic has had two shots of their COVID-19 vaccine.

### Who Will Know I Am in the Study?

Only my doctors and people who are involved in the study will know I am in it. When the study is finished, the doctors will write a report about what was learned. This report will not say my name or that I was in the study. My parents and I do not have to tell anyone I am in the study if we don't want to.

#### When Do I Have to Decide?

I have as much time as I want to decide to be part of the study. I have also been asked to talk about my decision with my parents.

#### Signatures

| If I put my name at the end of | of this form, | it means that I agree to be in the st | udy. |
|---|---|---|---|
| Participant's Signature | | Printed name | Date |
| Signature of Person Obtaining | Role | Printed name | <br>Date |